CLINICAL TRIAL: NCT06660966
Title: Comparison of the Effectiveness of M TAPA Block and ESP Block in Laparoscopic Cholecystectomy
Brief Title: Comparison of M-TAPA Block and ESP Block İn Laparoscopic Cholesystektomy
Acronym: MTAPA and ESP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Muharrem Baturu, Asisstant Prof. Dr, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANST01
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Postoperative Analgesia
Keywords: laparoscopic cholecystectomy; MTAPA block; ESP block; postoperative analgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group M (Active Comparator): M TAPA applied group
  Interventions: Procedure: M TAPA block
- Group E (Active Comparator): ESB applied Group
  Interventions: Procedure: ESP block group

INTERVENTIONS:
Procedure: M TAPA block — Grup M: The patients who underwent M-TAPA block were placed in the supine position. The right upper quadrant of the abdomen was cleaned with antiseptic solution. For the block procedure, 20-30 ml of 0.25% bupivacaine, 22G 8.5 cm stimuplex needle and 10-14 Hz high frequency USG were prepared for the procedure. The USG probe was determined in the costochondral area at the mid-clavicular line, and the internal and transversus abdominis muscles were determined. The needle was advanced with the in plane technique from cephalad to caudal, passing through the skin, subcutaneous, external and internal oblique muscles, respectively, and then over the transversus abdominis fascia. After the target was confirmed with 2 ml of saline, 0.3 mg / kg bupivacaine (20-30 ml) was administered.
  Arms: Group M
Procedure: ESP block group — In Group E, patients who were to undergo ESP block were placed in the lateral position with the right side up. The T8-T10 dorsal region was cleaned appropriately with antiseptic solution. For the block procedure, 20-30cc %0.25 bupivacaine, 22G 8.5cm stimuplex needle and 10-14Hz high frequency USG were prepared for the procedure.
  The USG probe is first determined in the sagittal direction, the spinous process of the T10 thoracic vertebra is then followed 1-2 cm above the transverse process, with the in plane technique, the skin, subcutaneous tissue and erector spina muscle are passed, the needle is touched to the transverse process and the target is confirmed with 2cc saline, then 20-30 cc (0.5 mg / kg bupivacaine) of local anesthetic is administered and the procedure is terminated.
  Arms: Group E

SUMMARY:
After cholecystectomy, modified-thoracoabdominal nerve block (M-TAPA) is a newly applied technique in upper abdominal surgery for postoperative analgesia. In recent years, block methods such as erector spina plane (ESP), paravertebral (PVB), transverses abdominis plane (TAP) have also been applied in these surgeries. MTAPA has been defined as a technique that is performed in the supine position and is easier to apply than the other mentioned blocks. In our study, we aimed to investigate the effectiveness of this block.

DETAILED DESCRIPTION:
After laparoscopic cholecystectomy, most patients experience moderate to severe pain, especially in the first 24 hours. The cause of the pain is the skin incision, the carbon dioxide insufflation given into the abdomen for laparoscopy, and the visceral peritoneum.

This pain that occurs in the postoperative period negatively affects the patient's early mobilization, wound healing, and patient comfort. While the toxic effects of nonsteroids used for pain control on the liver and kidneys are known, narcotic analgesics have side effects such as nausea, vomiting, and addiction. In recent years, trunk blocks have begun to be used frequently for pain control in abdominal surgery. Although blocks such as erector spina plane (ESP), paravertebral (PVB), and transverses abdominis plane (TAP) are frequently applied, there are differences in terms of their effectiveness and duration. On the other hand, it is important to give the patient a suitable position for the application.

Modified-thoracoabdominal nerve block (M-TAPA), which is applied especially in the supine position and is easier to apply compared to other blocks, has started to be applied as an alternative method.

In our study, we aimed to compare the effectiveness and duration of the MTAPA block compared to other trunk blocks such as ESP.

ELIGIBILITY:
Inclusion Criteria: ASAI-III , 18-70 yaş, elective surgery -

Exclusion Criteria: pregnancy, patient with emegency, patients allergic to local anesthetics, patient with coagülopaty, uncooperative, mentally retarded patients

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesia | postoperative 24 hours
  Numerical pain score below 3

CONTACTS AND LOCATIONS:
Locations (1):
- University of Gaziantep, Şehitkamil, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Altiparmak B, Korkmaz Toker M, Uysal AI, Turan M, Gumus Demirbilek S. The successful usage of modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) for analgesia of laparoscopic ventral hernia repair. J Clin Anesth. 2019 Nov;57:1-2. doi: 10.1016/j.jclinane.2019.02.016. Epub 2019 Mar 1. No abstract available. PMID 30831469
- [Background] Aikawa K, Tanaka N, Morimoto Y. Modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) provides a sufficient postoperative analgesia for laparoscopic sleeve gastrectomy. J Clin Anesth. 2020 Feb;59:44-45. doi: 10.1016/j.jclinane.2019.06.020. Epub 2019 Jun 15. No abstract available. PMID 31212124
- [Background] Bilge A, Basaran B, Et T, Korkusuz M, Yarimoglu R, Toprak H, Kumru N. Ultrasound-guided bilateral modified-thoracoabdominal nerve block through a perichondrial approach (M-TAPA) in patients undergoing laparoscopic cholecystectomy: a randomized double-blind controlled trial. BMC Anesthesiol. 2022 Oct 28;22(1):329. doi: 10.1186/s12871-022-01866-4. PMID 36307755
- See also: Related Info — https://bmcanesthesiol.biomedcentral.com/articles/10.1186/s12871-022-01866-4
- Available data/document: Statistical Analysis Plan — https://bmcanesthesiol.biomedcentral.com/articles/10.1186/s12871-022-01866-4 — The conformity of numerical data to normal distribution will be tested with the ShaphiroWilk test. Student t test will be used to compare variables that comply with normal distribution in 2 groups, and Mann Whitney U test will be used to compare variables that do not distribute normally in 2 groups. Relationships between categorical variables will be tested with the Chi-square test. Relationships between numerical variables will be tested with the correlation coefficient. SPSS 22.0 package program will be used in the analyses. A P value of less than 0.05 will be considered statistically significant.